CLINICAL TRIAL: NCT04483687
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Filgotinib in Subjects With Active Ankylosing Spondylitis Who Have an Inadequate Response to Biologic Disease-Modifying Antirheumatic Drug Therapy
Brief Title: Study to Evaluate the Efficacy and Safety of Filgotinib in Participants With Active Ankylosing Spondylitis Who Have an Inadequate Response to Biologic Disease-Modifying Antirheumatic Drug Therapy
Acronym: SEALION1-IR
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Development program terminated
Sponsor: Gilead Sciences (Industry)
Collaborators: Galapagos NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GS-US-433-5305; 2019-004298-24 (EudraCT Number)
Record Dates: First submitted 2020-07-20; First posted 2020-07-23 (Actual); Last update posted 2021-01-11 (Actual); Status verified 2021-01

CONDITIONS: Ankylosing Spondylitis
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — GLPG0634

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Filgotinib 200 mg (Main Study - Blinded) (Experimental): Participants will receive filgotinib 200 mg + placebo to match (PTM) filgotinib 100 mg for up to 16 weeks.
  Interventions: Drug: Filgotinib; Drug: Placebo to Match Filgotinib
- Filgotinib 100 mg (Main Study - Blinded) (Experimental): Participants will receive filgotinib 100 mg + PTM filgotinib 200 mg for up to 16 weeks.
  Interventions: Drug: Filgotinib; Drug: Placebo to Match Filgotinib
- Placebo (Main Study - Blinded) (Placebo Comparator): Participants will receive PTM filgotinib 200 mg + PTM filgotinib 100 mg for up to 16 weeks.
  Interventions: Drug: Placebo to Match Filgotinib
- Filgotinib 200 mg (LTE) (Experimental): Before study-wide unblinding, participants will receive filgotinib 200 mg + PTM filgotinib 100 mg.
  After study-wide unblinding, participants will receive filgotinib 200 mg.
  Interventions: Drug: Filgotinib; Drug: Placebo to Match Filgotinib
- Filgotinib 100 mg (LTE) (Experimental): Before study-wide unblinding, participants will receive filgotinib 100 mg + PTM filgotinib 200 mg.
  After study-wide unblinding, participants will receive filgotinib 100 mg.
  Interventions: Drug: Filgotinib; Drug: Placebo to Match Filgotinib

INTERVENTIONS:
Drug: Filgotinib — Tablets administered orally once daily
  Other Names: GS-6034; GLPG0634
  Arms: Filgotinib 100 mg (LTE); Filgotinib 100 mg (Main Study - Blinded); Filgotinib 200 mg (LTE); Filgotinib 200 mg (Main Study - Blinded)
Drug: Placebo to Match Filgotinib — Tablets administered orally once daily

SUMMARY:
The primary objective of this study is to evaluate the effect of filgotinib versus placebo on signs and symptoms of active ankylosing spondylitis (AS), evaluated by Assessment of SpondyloArthritis international Society 40% improvement (ASAS40) response at Week 16 in participants with active AS who have an inadequate response to biologic disease-modifying antirheumatic drug therapy.

DETAILED DESCRIPTION:
The study consists of 2 parts: Main Study (screening through Week 16) and Long-Term Extension (LTE) (up to 1.5 years after Week 16). Participants who permanently discontinue treatment in the Main Study will not be eligible for the Long-Term extension.

ELIGIBILITY:
Key Inclusion Criteria:

* Ambulatory male or female individuals who are ≥ 18 years of age (≥ 20 years of age in Japan) on the day of signing informed consent
* Have had inadequate response or intolerance to at least 1 and not more than 3 biologic disease-modifying antirheumatic drugs (bioDMARDs) administered for the treatment of ankylosing spondylitis (AS) or inflammatory arthritis
* Have an established diagnosis of radiographic axial spondyloarthritis (SpA)/ AS by a rheumatologist (or other specialist with expertise in diagnosing AS)
* Meet Assessment of SpondyloArthritis international Society (ASAS) classification criteria for axial SpA with radiographic sacroiliitis on imaging at screening as follows:

  * History of back pain ≥ 3 months and age at onset of back pain < 45 years, AND
  * Radiographic sacroiliitis Grade ≥ 2 bilaterally or Grade 3-4 unilaterally, AND
  * ≥ 1 SpA feature (refer to protocol; inflammatory back pain, arthritis, heel enthesitis, uveitis anterior, dactylitis, psoriasis, inflammatory bowel disease (IBD), good response to nonsteroidal anti-inflammatory drugs (NSAIDs), family history of SpA, historically positive human leukocyte antigen B27 (HLA-B27), elevated C-reactive protein (CRP))
* Have active AS at screening and Day 1 as defined by:

  * Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) ≥ 4, AND
  * Spinal pain ≥ 4 (based on BASDAI question 2)
* Have a history of inadequate response or intolerance to NSAIDs for the treatment of AS
* If using allowed conventional synthetic disease-modifying antirheumatic drugs (csDMARDs), NSAID, or corticosteroid therapy, must have been on stable doses (as outlined in protocol) prior to Day 1

Key Exclusion Criteria:

* Prior exposure to a Janus kinase (JAK) inhibitor > 2 doses
* Total ankylosis of the spine
* Any active/recent infection, as specified in the protocol
* Diagnosis of fibromyalgia
* Any musculoskeletal disorder other than AS that would interfere with assessment of study parameters, as per judgement of investigator

  * Note: Prior history of reactive or other types of inflammatory arthritis is permitted if there is documentation of change in diagnosis to AS or additional diagnosis of AS
* Any history of an inflammatory arthritis with onset age before 16 years old

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-12 (Estimated); Primary Completion 2023-01 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Proportion of Participants Who Achieve an Assessment of SpondyloArthritis international Society 40% Improvement (ASAS40) Response at Week 16 | Week 16
  The ASAS40 calculation involves the analysis of 4 domains: participant's global assessment of disease activity, spinal pain (derived from the spinal pain questionnaire), function (derived from Bath Ankylosing Spondylitis Functional Index (BASFI) score), and inflammation (derived from morning stiffness questions from Bath Ankylosing Spondylitis Disease Activity Index (BASDAI)). The ASAS40 is achieved if there is an improvement of ≥ 40% and ≥ 2 units in at least 3 domains on a scale of 10 with no worsening in the remaining domain.

SECONDARY OUTCOMES:
Proportion of Participants Who Achieve an ASAS40 Response | Up to Week 12
  The ASAS40 calculation involves the analysis of 4 domains: participant's global assessment of disease activity, spinal pain (derived from the spinal pain questionnaire), function (derived from BASFI score), and inflammation (derived from morning stiffness questions from BASDAI). The ASAS40 is achieved if there is an improvement of ≥ 40% and ≥ 2 units in at least 3 domains on a scale of 10 with no worsening in the remaining domain.
Proportion of Participants Who Achieve an Assessment of SpondyloArthritis international Society 20% Improvement (ASAS20) Response | Up to Week 16
  The ASAS20 calculation involves the analysis of 4 domains: participant's global assessment of disease activity, spinal pain (derived from the spinal pain questionnaire), function (derived from BASFI score), and inflammation (derived from morning stiffness questions from BASDAI).The ASAS20 is achieved if there is an improvement of ≥ 20% and ≥ 1 units in at least 3 domains on a scale of 10 with no worsening of ≥ 20% and ≥ 1 unit in the remaining domain.
Proportion of Participants who achieve Ankylosing Spondylitis Disease Activity Score (ASDAS) Low Disease Activity (LDA) (ie, ASDAS < 2.1) at Week 16 | Week 16
  ASDAS is a composite score of 5 domains: total back pain, peripheral pain and/or swelling, duration of morning stiffness (derived from BASDAI questionnaire), participant's global assessment of disease activity, and serum high-sensitivity C-reactive protein (hsCRP). The ASDAS has a continuous scale from 0 with no defined upper end. A lower score indicate lower disease activity. ASDAS LDA is achieved when ASDAS < 2.1.
Proportion of Participants Who Achieve an ASAS 5/6 Response | Up to Week 16
  The ASAS 5/6 is achieved when at least 20% improvement in at least 5 out of 6 domains. The 6 domains to use are: participant's global assessment of disease activity, spinal pain (derived from the spinal pain questionnaire), function (derived from BASFI score), inflammation (derived from morning stiffness questions from BASDAI), lateral spinal flexion (Bath Ankylosing Spondylitis Metrology Index (BASMI) question 1), and hsCRP.
Change from Baseline in the Individual Components of the ASAS Core Set | Baseline and up to Week 16
  ASAS core set consists of 6 assessment domains: (1) participant's global assessment of disease activity, (2) spinal pain (derived from the spinal pain questionnaire), (3) function (derived from BASFI score), (4) inflammation (derived from morning stiffness questions from BASDAI), (5) hsCRP, (for these 5 domains, a lower score indicate lower disease activity) and (6) lateral spinal flexion (BASMI question 1) (for this 6th domain; a higher score indicate lower disease activity).
Proportion of Participants Who Achieve a Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) 50% Improvement Response | Up to Week 16
  BASDAI consists of 6 items asking participants to report their fatigue, spinal pain, peripheral arthritis, enthesitis, intensity, and duration of morning stiffness during the past week on a 0 to 10 numeric rating scale. The total score ranges 0-10; scores of 4 or greater suggest suboptimal control of disease. BASDAI 50% improvement is achieved when a decrease in BASDAI versus baseline by at least 50%.
Change From Baseline in ASDAS | Baseline and up to Week 16
  ASDAS is a composite score of 5 domains: total back pain, peripheral pain and/or swelling, duration of morning stiffness (derived from BASDAI questionnaire), participant's global assessment of disease activity, and hsCRP. The ASDAS has a continuous scale from 0 with no defined upper end. A lower score indicates lower disease activity.
Change From Baseline in BASDAI | Baseline and up to Week 16
  BASDAI consists of 6 items asking participants to report their fatigue, spinal pain, peripheral arthritis, enthesitis, intensity, and duration of morning stiffness during the past week on a 0 to 10 numeric rating scale. The total score ranges 0-10; scores of 4 or greater suggest suboptimal control of disease.
Change From Baseline in Bath Ankylosing Spondylitis Functional Index (BASFI) | Baseline and up to Week 16
  The BASFI evaluates physical function in AS. The instrument consists of 10 items, rated on a 0 to 10 numeric rating scale (NRS), where 0 represents "easy" and 10 represents "impossible." Among the 10 items, 8 items evaluate basic activities of daily living (putting on socks, bending, reaching up, 2 items on getting up, standing, climbing steps, and looking over shoulder) and 2 items assess participants' ability to cope with everyday life (physically demanding activities and full day's activities). The total score ranges 0-10, and the higher the score, the higher the functional impairment.
Change From Baseline in Bath Ankylosing Spondylitis Metrology Index (BASMI) (Linear Score) | Baseline and up to Week 16
  The BASMI combines 5 measures: lateral spinal flexion, tragus-to-wall distance, lumbar flexion (modified Schober index), maximal intermalleolar distance, and cervical rotation. The BASMI will be scored using a linear function that will quantify the mobility of the axial skeleton and allow for objective assessment of clinically significant changes in spinal movement. The total score ranges 0-10, and the higher the score, the more severe the participant's limitation on movement.
Change From Baseline in Chest Expansion | Baseline and up to Week 16
  Chest expansion will be measured during maximal inspiration and maximal forced expiration at the fourth intercostal space.
Change From Baseline in Occiput-to-wall Distance | Baseline and up to Week 16
  Occiput-to-wall distance is measured twice with the participant's heels and back rested against the wall. The chin should be at usual carrying level and the participant takes maximal effort to touch the head against the wall. The distance between the occiput and the wall is assessed and the better of the 2 assessments is to be reported.
Change From Baseline in Maastricht Ankylosing Spondylitis Enthesitis Score (MASES), in Participants With Enthesitis at Baseline | Baseline and up to Week 16
  MASES is based on enthesitis grading of 13 body sites. The MASES is the sum of all site scores and ranges from 0-13. The higher the score, the higher the presence of enthesitis.
Change From Baseline in Ankylosing Spondylitis Quality of Life (ASQoL) | Baseline and up to Week 16
  The ASQoL assesses health-related quality of life in AS participants. The questionnaire consists of 18 yes/no questions. A single point will be assigned for each "yes" response, resulting in a total score between 0 and 18, with lower scores indicating a better quality of life.
Change From Baseline in Assessment of SpondyloArthritis international Society Health Index (ASAS HI) | Baseline and up to Week 16
  The ASAS HI is a 17-item patient-reported outcome measure to assess the impact of interventions for spondyloarthritis (SpA), including axial SpA. Each item consists of a question with a binary response of either "I agree" (scored as 1) or "I do not agree" (scored as 0). The scoring is performed by summing the number of "yes" answers. The total sum of the ASAS HI ranges 0-17, with a lower score indicating a better health status.
Change From Baseline in Physical Component Summary (PCS) Score of the 36-Item Short-Form Survey (SF-36) Version 2 | Baseline and up to Week 16
  The SF-36 Version 2 is a health-related survey that assesses participant's quality of life and consists of 36 questions covering 8 health domains: physical functioning, bodily pain, role limitations due to physical problems and emotional problems, general health perceptions, mental health, social functioning, vitality, and 2 component scores (Mental Component Summary (MCS) score and PCS). MCS consists of social functioning, vitality, mental health, and role-emotional. PCS consists of physical functioning, bodily pain, role-physical, and general health perceptions. Each domain will be scored by summing the individual items and transforming the scores into a 0 to 100 scale with higher scores indicating better health status or functioning.
Change From Baseline in Mental Component Summary (MCS) Score of the SF-36 Version 2 | Baseline and up to Week 16
  The SF-36 Version 2 is a health-related survey that assesses participant's quality of life and consists of 36 questions covering 8 health domains: physical functioning, bodily pain, role limitations due to physical problems and emotional problems, general health perceptions, mental health, social functioning, vitality, and 2 component scores (MCS and PCS). MCS consists of social functioning, vitality, mental health, and role-emotional. PCS consists of physical functioning, bodily pain, role-physical, and general health perceptions. Each domain will be scored by summing the individual items and transforming the scores into a 0 to 100 scale with higher scores indicating better health status or functioning.
Change from Baseline in Functional Assessment of Chronic Illness Therapy - Fatigue Scale (FACIT-Fatigue) | Baseline and up to Week 16
  The FACIT-Fatigue measures an individual's level of fatigue during their usual daily activities during the past week. It consists of 13 questions on a 5-point Likert scale, with 0 indicating "not at all" and 4 indicating "very much". Negatively stated items are reversed and the total score ranges 0-52. Low scores indicate more severe fatigue than high scores.
Change From Baseline in Work Productivity and Activity Impairment for Ankylosing Spondylitis (WPAI-AS) | Baseline and up to Week 16
  The WPAI-AS is a questionnaire developed to measure impairments in work activities in participants with AS. The questionnaire consists of 6 questions (currently employed, work time missed due to AS, work time missed due to other reasons, hours actually worked, degree AS affected productivity while working [0-10 NRS; with 0 indicating no effect and 10 indicating AS completely prevented the participant from working], and degree AS affected productivity in regular unpaid activities [0-10 NRS; with 0 indicating no effect and 10 indicating AS completely prevented the participant's daily activities]). The recall period for questions 2 through 6 is 7 days.
  Four main outcomes (expressed in percentages) can be obtained from the WPAI-AS: percentage of work time missed due to AS, percentage of impairment due to AS, percentage of overall work impairment due to AS, and percentage of activity impairment due to AS. Higher numbers indicate greater impairment and less productivity.
Change From Baseline in EuroQol 5 Dimensions 5 Levels (EQ-5D-5L) | Baseline and up to Week 16
  The EQ-5D-5L is a standard measure of health-related quality of life. The tool consists of the EQ-5D-5L descriptive system and the EQ visual analogue scale (VAS). The descriptive part comprises 5 dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression). Each of these 5 dimensions has 5 levels (no problem, slight problems, moderate problems, severe problems, and extreme problems). Results for each of the 5 dimensions are combined into a 5-digit number to describe the participant's health state. The VAS records the participant's health on a 0-100 mm VAS scale, with 0 indicating "the worst health you can imagine" and 100 indicating "the best health you can imagine." Higher scores of EQ VAS indicate better health.

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences

IPD SHARING:
Plan to Share IPD: No